CLINICAL TRIAL: NCT03807479
Title: Phase 2 Clinical Trial With Ponatinib as a Second Line Therapy for Patients With Chronic Myeloid Leukemia in Chronic Phase Resistant or Intolerant to Prior First Line Tyrosine Kinase Inhibitor Treatment
Brief Title: Study in Patients With Chronic Leukemia
Acronym: PONS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: less recruting
Sponsor: GWT-TUD GmbH (Other)
Collaborators: Incyte Biosciences International Sàrl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PONS_11272
Record Dates: First submitted 2018-11-07; First posted 2019-01-17 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-09

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
Keywords: CP-CML; CML in chronic phase; Chronic Myelogenous Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ponatinib (Experimental): Patients in this treatment arm receive Ponatinib: starting dose 30 mg once-daily. Doses may be increased in case of inappropriate response and reduced to manage drug-related adverse events (AEs) and may be re-escalated once events resolve.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — 2 film-coated tablets à 15mg for oral administration on a daily basis
  Other Names: Iclusig

SUMMARY:
This study will include patients suffering from chronic myeloid leukemia (CP-CML), who were treated with tyrosine kinase inhibitor (TKI, a substance that blocks the action of enzymes) in a previous therapy but which has not been effective. Patients will be treated with Ponatinib 30 mg in in this study. The aim of the study is to evaluate the safety and efficacy of Ponatinib as a second line treatment in patients failing or not tolerating first line therapy with any other approved TKIs. It is expected that Ponatinib, due to its efficacy, may be more effective as second line therapy than other approved TKIs and lead to improved overall survival. The effect will be determined by the molecular response rate (MMR) as the primary objective after 12 months of treatment. The safety of the drug will be evaluated on the basis if routine medical and laboratory examinations.

DETAILED DESCRIPTION:
Despite significant progress in the treatment of patients with chronic phase CML, there is still need to further optimize therapy to reach the goal of disease eradication for almost all patients. In case of imatinib failure, dasatinib and nilotinib are effective treatment options after an individualized treatment selection. Although MMR rates of around 30% after 2 years of therapy are a significant achievement, options that may improve response rates in depth are still desirable. Ponatinib is a third generation TKI with very high anti-clonal activity in all CML phases. Moreover, it also eradicates most of the known and problematic mutations and only very few (compound) mutations may induce ponatinib-resistance.

Based on its favourable target spectrum, it is expected that Ponatinib may be more effective than 2nd line dasatinib or nilotinib in achieving early (i.e., at 6 months) cytogenetic and molecular responses in patients after inappropriate response to imatinib, and more effective as 2nd line treatment after failure of initial treatment with dasatinib or nilotinib than a cross-over between the 2nd generation TKIs. The basic hypothesis underlying therapeutic programs in CML is to be able to achieve meaningful and long-lasting suppression of the Philadelphia chromosome and breakpoint cluster region-abelson fusion gen (BCR-ABL). Complete cytogenetic responses have been associated with improved survival in CML, while major molecular responses are associated with improved event-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years old
2. Diagnosis of Ph-positive (by cytogenetics) or BCR-ABL-positive (by PCR) CP-CML
3. Patients should have demonstrated to have

   * a failure of a prior 1st line TKI treatment with either imatinib, dasatinib or nilotinib. Failure is defined as per European LeukemiaNet (ELN) recommendations:

     * Less than Complete Hematologic Response (CHR) and/or Ph+ > 95% at or beyond 3 months
     * No cytogenetic response (Ph+>35%) and/or Abelson murine leukemia viral oncogene homolog 1 (BCR-ABL1) >10% at or beyond 6 months
     * BCR-ABL (on international scale) >1% and/or PH+ >0%
     * Less than MMR at or beyond 18 months
     * Loss of response or development of mutations or other clonal chromosomal abnormalities at any time during the first line TKI treatment
   * or intolerance to prior TKI treatment defined as grade 3 or 4 toxicity, or persistent grade 2 toxicity despite optimal management including dose adjustment, or in a patient where dose reductions are considered to be not in the patient's best interest to obtain an adequate response. Intolerant patients should not have achieved or have lost major molecular response at the time of enrollment
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

Exclusion Criteria:

1. Any 1st line anti-CML treatment other than TKI (apart from therapy with hydroxyurea)
2. Any 2nd line therapy with a tyrosine kinase inhibitor (>1 European Medicines Agency (EMA) approved TKI for CML, or any investigational non EMA-approved TKI)
3. Concurrent participation in any other clinical trial involving another investigational drug within 4 weeks prior to enrollment and throughout participation in PONS-Study
4. New York Heart Association (NYHA) cardiac class 3-4 heart disease
5. Cardiac Symptoms within the past 12 months prior recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Major Molecular Response (MMR) of treatment | by 12 moths
  To estimate the proportion of CP-CML patients with tyrosine kinase inhibitor (TKI)-resistance or intolerance to first line therapy with TKI, attaining MMR by 12 months of treatment with second line Ponatinib therapy.

SECONDARY OUTCOMES:
Time to toxicity | up to 24 months
  To evaluate the toxicity profile of ponatinib in patients with CML in chronic phase after one TKI failure toxicities will be followed up at each visit during the treatment phase and will be assessed using CTCAE v.5.0. Type of toxicity (hematologic or non-hematologic) along with the grading will be followed up on.
Time to response | at 3, 6, 9, 12, 18 and 24 months
  To estimate the time to CCyR, MMR, MCyR and MR4 for patients treated with Ponatinib as second line therapy for CP-CML (chronic phase-chronic myelogenous leukemia).
Durations of response | at 3, 6, 9, 12, 18 and 24 month
  To evaluate the duration of hematologic, cytogenetic and molecular response to Ponatinib after one TKI failure.
Occurrence of BCR-ABL-mutations | at 3, 6, 9, 12, 18 and 24 months
  To evaluate the occurrence of BCR-ABL-mutations in patients with failure of Ponatinib 2nd line therapy.
Time to progression | at 3, 6, 9, 12, 18 and 24 months
  To define the time to progression for patients with CML in chronic phase treated with Ponatinib after one TKI failure.
Time to overall survival | at 3, 6, 9, 12, 18 and 24 month
  To define the time to overall survival for patients with CML in chronic phase treated with Ponatinib after one TKI failure.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp le Coutre, Prof., Principal Investigator — Charité Berlin - Department of Hematology, Oncology and Tumor Immunology
Locations (10):
- Germany (10):
  - University Hospital, Halle, Saxony-Anhalt
  - University Hospital RWTH Aachen,Clinic for Hematology, Oncology, Hemostaseology and Stem Cell Transplantation, Medical Department IV, Aachen
  - Charité University Medicine Berlin - Medical Clinic, Department of Hematology, Oncology and Tumor Immunology, Berlin
  - University Hospital Essen gGmbH, Westdeutsches Tumorzentrum; Internal Medicine (Tumor Research), Essen
  - University Medicine Greifswald, Clinic and Policlinic - Internal Medicine C - Hematology and Oncology, Greifswald
  - Asklepios Clinic St. Georg - Department of Oncology, Section Hematology, Hamburg
  - University Hospital Mannheim GmbH, III. Medical Clinic for Hematology and Oncology, Mannheim
  - Clinic for Hematologie, Marburg
  - UKRUB University Hospital of Ruhr-University Bochum, Clinic for Hematology and Oncology, Minden
  - University Hospital Ulm - Department for internal medicine III, Ulm

IPD SHARING:
Plan to Share IPD: No